CLINICAL TRIAL: NCT01007617
Title: Evaluation of Low-energy Laser Therapy for Prevention and Reduction of Severity of Oral Mucositis in Children "Mucositis Laser 1"
Brief Title: Low-energy Laser Therapy for Prevention of Oral Mucositis in Children
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre Régional de Cancérologie et Thérapie Cellulaire Pédiatrique, CHU de Clermont-Ferrand (Unknown); Faculté de chirurgie dentaire, Clermont-Ferrand (Unknown); Centre de Pharmacologie Clinique, INSERM CIC 501 (Unknown); Laboratoire des Matériaux Inorganiques, ESA CNRS 6002 et ENSCCF, Université Blaise-Pascal, Aubière (Unknown)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0060
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Oral Mucositis
Keywords: Children; Cancer; Mucositis; Laser; Prevention; Chemotherapy; Children with malignancies receiving chemotherapy and/or radiotherapy inducing severe mucositis
MeSH Terms: conditions — Stomatitis; Neoplasms; Mucositis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Device: LLLT :low level laser therapy — The patients will be randomized in 2 groups according to the delivered dose: 2 J/cm2/d or 8 J/cm2/d.
  Main evaluation criteria: mucositis maximal intensity (WHO scale).
  Secondary evaluation criteria: mucositis duration, mucositis survival free, pain, opioid treatment, hospitalization, fever and infection, nutrition.

SUMMARY:
Oral mucositis represents a major complication of cytotoxic chemotherapy among cancer in children. Low-power laser therapy (LPLT) has been used to reduce the incidence of oral mucositis in patients who are receiving high-dose chemotherapy. The aim of this study is to compare two preventives energies delivered of LPLT to oral mucosa in decreasing the severity of mucositis in children.

DETAILED DESCRIPTION:
Mucositis is one of the main complications of cytotoxic chemotherapy and total body irradiation in children cancers. Local and systemic treatments are not efficiency or limited by side effects, (particularly for opioid). Two randomized recent studies in adult have showed the efficiency of LPLT (wavelength 650nm at the intensity of 4J/cm²) in prevention of severe mucositis. In pediatrics patient, only one randomized study was performed to the same intensity of 4J/cm² but with a wavelength of 732nm, and did not show the evidence of profit. In theory, tissues absorption level of laser is similar at 650 and 900nm but lower around 700nm. Procedure was very well tolerated by children; the main limiting factor is the deadline directly proportional to intensity delivered.

The aim of our study is to compare two preventives energies (2J/cm² or 8 J/cm²) daily delivered of LPLT to oral mucosa in decreasing the severity of mucositis in children. Placebo study was not possible to our opinion and we preferred to compare two intensity of LPLT for three reasons : being given the sensation of heat generated by the treatment, a true placebo is difficult to obtain; considering the difficulties proceeding to large-sized clinical trials in this population, it seems to us necessary to end quickly in an optimal protocol; the main inconvenience of LPLT is the duration of the sessions, so in case of negative result, our study will generate data allowing not to realize useless too long sessions.

It's a prospective controlled study, randomized in double blind phase II, in one center. All the patients will receive LPLT (GaAlAs, wavelength 980nm) daily of the 1st in the 5th day of cytotoxic treatment. The patients will be randomized in 2 groups according to the delivered dose: 2 J/cm2/d or 8 J/cm2/d.

Main evaluation criteria: mucositis maximal intensity (WHO scale) Secondary evaluation criteria: mucositis duration, mucositis survival free, pain, opioid treatment, hospitalization, fever and infection, nutrition.

Expected clinical effects: improvement of the children's comfort; dissemination of the technique in the other oncology pediatric centers

ELIGIBILITY:
Inclusion Criteria:

* 0 at 18 years
* patients receiving therapy with agents likely to cause severe mucositis (grade 3 or 4)
* Patients who had developed severe mucositis previously in any chemotherapy, and receiving the same.
* Healthy oral mucosa
* informed consent

Exclusion Criteria:

* - Infection active and proved, viral, bacterial or fungal oral cavity
* Malignant pathology in the oral cavity
* Preliminary local irradiation of the oral cavity
* Simultaneous treatment by an agent of prevention or treatment of mucositis in investigation
* Inclusion in a protocol with oral mucositis as one of the assessment criteria
* Absence of consent lit by parents or child

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Mucositis scale - World Health Organization (WHO) | after delivering a dose of 2 J/cm2/d

SECONDARY OUTCOMES:
Mucositis period | after delivering a dose of 8 J/cm2/d
Mucositis free survival | after delivering a dose of 8 J/cm2/d
Pain intensity | after delivering a dose of 8 J/cm2/d
Morphinic administration | after delivering a dose of 8 J/cm2/d
Duration of hospitalisation | after delivering a dose of 8 J/cm2/d
Febrile neutropenia | after delivering a dose of 8 J/cm2/d
Duration of parenteral nutrition | after delivering a dose of 8 J/cm2/d
Psychological impact | after delivering a dose of 8 J/cm2/d

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MERLIN, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France